CLINICAL TRIAL: NCT06291142
Title: NIHR i4i 2: Early Diagnosis of Systemic Sclerosis in the General Rheumatology Clinic - Pilot Image Acquisition Study
Brief Title: Early Diagnosis of SSc in the General Rheumatology Clinic - Pilot
Status: Completed | Type: Observational
Sponsor: University of Manchester (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); Royal Bolton Hospital NHS Foundation Trust (Other); Alder Hey Children's NHS Foundation Trust (Other); University Hospitals of Morecambe Bay NHS Trust (Other); Stockport NHS Foundation Trust (Other); Medway NHS Foundation Trust (Other); Northern Care Alliance NHS Foundation Trust (Other); Royal Free Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: R129030; IRAS 315004 (Other: IRAS)
Record Dates: First submitted 2024-02-26; First posted 2024-03-04 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2024-02

CONDITIONS: Systemic Sclerosis; Raynaud Phenomenon
Keywords: Raynaud's; Systemic Sclerosis Spectrum Disorder; Artificial Intelligence; Imaging; Capillaroscopy; Scleroderma
MeSH Terms: conditions — Scleroderma, Systemic; Raynaud Disease; Scleroderma, Diffuse

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patient Participants: Patients with an SSc spectrum disorder, and healthy controls (objective 3)
  Interventions: Device: Observation - Nailfold capillaroscopy
- Healthcare Professional Participants: Healthcare Professionals taking part in the qualitative element of the study
  Interventions: Device: Observation - Nailfold capillaroscopy

INTERVENTIONS:
Device: Observation - Nailfold capillaroscopy — Nailfold capillaroscopy examination

SUMMARY:
The goal of this observational pilot data acquisition study is to establish if target users can obtain diagnostic quality images in the clinic, from participants with Systemic Sclerosis (SSc), and SSc spectrum conditions. The main questions it aims to answer are:

* Can a range of healthcare professionals, including non-specialists, use the capillaroscopy image acquisition system to take high quality images that can be used to create a clinical report?
* Can the investigators collect user and patient feedback on the usability of the capillaroscopy system, to help develop the software and to develop the clinical report
* Which microscope light source, from four different light wavelengths is better to see the blood vessels in skin with more melanin content.

Participants will be asked to attend a single clinic visit where they will undergo a brief, non-invasive nailfold capillaroscopy examination, using the software-guided capillaroscopy system.

Participants and rheumatology healthcare professionals will be invited to take part in one or more focus groups and interviews, to collect feedback and to contribute to the development of the image acquisition software and the clinical report.

DETAILED DESCRIPTION:
Systemic sclerosis (SSc) is a painful, disabling disease affecting around 20,000 people in the UK. Symptoms include painful ulcers on the fingers and toes, sometimes requiring amputation, and life-threatening internal organ damage. The first symptom of SSc is usually Raynaud's phenomenon - white, painful fingers in the cold - though around 5% of otherwise healthy individuals also experience Raynaud's. The National Institute for Health and Care Excellence (NICE) recommends that GPs should refer patients with Raynaud's to a general rheumatology clinic for assessment. When a patient is referred for assessment, using nailfold capillaroscopy to find vessel abnormalities caused by SSc is recognised internationally as key to early diagnosis. Despite this, it is not used in most rheumatology clinics, because it requires expensive equipment and specialised skill. When capillaroscopy is not available, diagnosis is often delayed, which can have serious consequences for patients.

The research team will develop an artificial intelligence (AI) system that helps rheumatology clinics diagnose SSc as early as possible. The system will use nailfold capillaroscopy images of the small blood vessels at the base of the fingernails and digital technology to find changes due to disease. In a previous study has shown that, in expert hands, capillaroscopy images good enough to diagnose SSc can be obtained using a commercially available, hand-held microscope. The investigators have also developed AI image analysis software that finds capillary abnormalities very reliably.

This study will establish if target users can acquire diagnostic-quality images in clinic and provide feedback to inform technology refinement. Images will be acquired using version one of our software from 105 patients across seven centres in England. The investigators will also run focus groups and interviews to gain qualitative input from users and patients to assess usability of the system. The results of this study will contribute to the development of a complete system suitable for use by non-specialists.

ELIGIBILITY:
Inclusion Criteria:

Image Acquisition:

* Children (aged between 6-17 years) and adults (aged 18 years and above) with Raynaud's phenomenon or a SSc- spectrum disorder.

Qualitative aspect:

* Rheumatologists, vascular technicians, specialist nurses, or similar rheumatology trained professionals
* Patients with Raynaud's phenomenon and/or a SSc-spectrum disorder.
* Adults ages 18 years and over.

Exclusion Criteria:

* (Patients; image acquisition and skin tone study). Diabetes
* (Healthy controls). Requirement for vasoactive therapies
* (Healthy controls). Any condition known to affect the vasculature e.g. unregulated hypertension
* (All groups). Any disorder limiting the ability to provide informed consent or to comply with study requirements.

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be identified by a review of patient medical records, or patients who present at a clinic appointment.
  Healthy controls (only applicable to the skin tone study at Salford Royal) will be identified via a database of previous volunteers, and via advertisements.
  Rheumatologists, vascular technicians, specialist nurses and other associated professionals required to take part in the focus groups and interviews will likely be those from each of the collaborating sites. They will be informed of the opportunity to take part during meetings with the research team and will be sent a participant information sheet via email.
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2023-11-22 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Pilot Image Acquisition | 11 months
  A set of nailfold capillaroscopy images from each participant

SECONDARY OUTCOMES:
Qualitative Feedback | 11 months
  A set of qualitative feedback data collected from patient participants and HCPs
Skin tone sub-study data set | 11 months
  A set of nailfold capillaroscopy images collected from participants from a range of Fitzpatrick Skin Scores, using 4 different light wavelength cameras

CONTACTS AND LOCATIONS:
Overall Officials: Ariane E Herrick, MD, FRCP, Principal Investigator — The University of Manchester
Locations (1):
- Northern Care Alliance NHS Foundation Trust, Salford, Salford, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Herrick AL, Berks M, Taylor CJ. Quantitative nailfold capillaroscopy-update and possible next steps. Rheumatology (Oxford). 2021 May 14;60(5):2054-2065. doi: 10.1093/rheumatology/keab006. PMID 33493310